CLINICAL TRIAL: NCT04170205
Title: Retrospective Study of Causes Associated With Small Fiber Neuropathies.
Brief Title: Causes Associated With Small Fiber Neuropathy (SFN).
Acronym: EtioNPF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19. 0218 (EtioNPF)
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Small fiber neuropathy (SFN) is an injury of cutaneous nerve fibers, mainly by a decrease in their density within the cutaneous tissue. The symptomatology associated with this SFN is broad with symptoms that are essentially sensory, but also autonomic. The etiologies of SFN are numerous (diabetes, drug, infectious, immunological...) and clinically non-specific, justifying a broad etiological assessment. The appearance of staged skin biopsies in the SFN balance sheet has greatly helped to improve diagnosis.

Despite this, a significant part of SFN remains without associated etiology and is considered idiopathic.

As the distribution of the different causes of SFN remains a missing data to date, the completion of this cohort study by one of the SFN reference centres should make it possible to establish the prevalence of SFN causes over a large population.

Only patients with clinical symptoms that may be related to SFN and who have been sampled for SFN, positive or not, will be eligible for recruitment.

The result of the anatomopathological sampling will allow patients to be separated into two groups, with or without SFN.

The main judgement criteria will be the prevalence of etiologies associated with SFN: diabetes, medication, systemic lupus erythematosus, Gougerot-Sjögren syndrome, amylosis, dysthyroidism, alcoholism, vitamin B12 deficiency, HIV infection, hepatitis C, paraneoplastic syndrome, hereditary disease (Fabry disease, Friedreich ataxia,...), idiopathic, others.

ELIGIBILITY:
Inclusion Criteria:

* Age of majority (>18 years old)
* Clinically managed patient at Brest University Hospital
* Patient who had a skin biopsy with anatomopathological examination for SFN performed at the University Hospital of Brest

Exclusion Criteria:

* Under age of majority (<18 years old)
* Patient not followed at Brest University Hospital
* Refusal to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical symptomatology in favour of SFN who have been subjected to skin histological examination for SFN
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of etiologies associated with SFN | 1 year
  Source population will be patients with symptoms that may be related to SFN, who have performed a biopsy for SFN.
  Patient will be considered to have SFN if he or she has a decrease in intra-epidermal distal density at nerve endings below the 5th percentile and at least one clinical sign in favour of small fibre neuropathy.
  Clinical signs in favour of SFN are as follows :
  Sensitive symptoms: burns, stings, numbness, tingling, hot/cold sensations, electric shocks, hyperesthesia, allodynia, intolerance of bed sheets, pruritus, restless legs.
  Vegetative symptoms: erectile disorders, dry syndrome, sweating, hot flashes, vertigo/discomfort (orthostatic hypotension), digestive and/or urinary disorders, resting tachycardia, palpitations
  Vascular symptoms: erythromelalgia, acrosyndrome

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.